CLINICAL TRIAL: NCT02402491
Title: Twelve Versus 24 Months of Dual Antiplatelet Therapy in Patients With Percutaneous Coronary Intervention for In-stent Restenosis
Brief Title: Twelve vs 24 Months of Dual Antiplatelet Therapy in Patients With Coronary Revascularization for In-stent Restenosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, professor of cardiology, vice president of Beijing Anzhen Hospital, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISR-DAPT
Record Dates: First submitted 2015-03-23; First posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Dual Antiplatelet Treatment; In-Stent Restenosis
MeSH Terms: interventions — Purinergic P2Y Receptor Antagonists; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 24 months of P2Y12 receptor antagonist (Active Comparator): Receive 24 months of dual antiplatelet therapy (with a P2Y12 receptor antagonist in addition to aspirin) after index procedure. All subjects receive aspirin for the duration of study.
  Interventions: Drug: 24 months of P2Y12 receptor antagonist; Drug: Aspirin
- 12 months of P2Y12 receptor antagonist (Placebo Comparator): Receive 12 months of dual antiplatelet therapy (with a P2Y12 receptor antagonist in addition to aspirin) after index procedure. All subjects receive aspirin for the duration of study.
  Interventions: Drug: 12 months of P2Y12 receptor antagonist; Drug: Aspirin

INTERVENTIONS:
Drug: 12 months of P2Y12 receptor antagonist — All subjects will be received 12 months of dual antiplatelet therapy with a P2Y12 receptor antagonist (clopidogrel/prasugrel/ticagrelor) in addition to aspirin.
  Arms: 12 months of P2Y12 receptor antagonist
Drug: 24 months of P2Y12 receptor antagonist — All subjects will be received 24 months of dual antiplatelet therapy with a P2Y12 receptor antagonist (clopidogrel/prasugrel/ticagrelor) in addition to aspirin.
  Arms: 24 months of P2Y12 receptor antagonist
Drug: Aspirin — The maintenance dose of aspirin is 100 mg daily, to be taken indefinitely.

SUMMARY:
Patients undergoing the percutaneous coronary intervention (PCI) for in-stent restenosis (ISR) are enrolled. All patients will be randomized to receive either 12 months or 24 months of dual antiplatelet therapy with a P2Y12 receptor antagonist in addition to aspirin, all patients continue receiving aspirin indefinitely. The primary efficacy end points of this study are the incidence of a composite end point including all cause deaths, myocardial infarction, the incidence of Academic Research Consortium defined definite or probable stent thrombosis and stroke (MACCE) at 24 months. The primary safety end point is the incidence of GUSTO moderate or severe bleeding.

DETAILED DESCRIPTION:
The ISR-DAPT Study is a multicenter, randomized controlled trial that will enroll 1000 subjects treated with percutaneous coronary intervention (PCI) for in-stent restenosis. All patients will be randomized to receive either 12 months or 24 months of dual antiplatelet therapy with a P2Y12 receptor antagonist in addition to aspirin after index procedure. All patients continue receiving aspirin indefinitely. The primary efficacy end points of this study are the incidence of a composite end point including all cause deaths, myocardial infarction, the incidence of Academic Research Consortium defined definite or probable stent thrombosis and stroke (MACCE) at 24 months. The primary safety end point is the incidence of GUSTO moderate or severe bleeding at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-80 years of age
* Undergoing percutaneous intervention with stent deployment for the treatment of in-stent restenosis

Exclusion Criteria:

* Pregnant women
* Planned surgery necessitating discontinuation of antiplatelet therapy within the 24 months after enrollment
* Current medical condition with a life expectancy of <2 years
* Concurrent enrollment in another device or drug study whose protocol specifically rules out concurrent enrollment
* Subjects on warfarin or similar anticoagulant therapy
* Subjects with hypersensitivity or allergies to one of the drugs
* Subjects unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
MACCE | 24 months
  Incidence of a composite end point including all cause deaths, myocardial infarction, the incidence of Academic Research Consortium defined definite or probable stent thrombosis and stroke (MACCE) at 24 months.

SECONDARY OUTCOMES:
Safety end point assessed by incidence of GUSTO moderate or severe bleeding. | 24 months
  Specifically, bleeding complications are classified as severe if they are intracerebral or if they result in substantial hemodynamic compromise requiring treatment. Moderate bleeding is defined by the need for transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, MD, PhD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China